CLINICAL TRIAL: NCT02062307
Title: Osteoprotegerin, Fibroblast Growth Factor 23 and Vitamin D3 Levels in Male Patients With Hypogonadism
Brief Title: Bone Mineral Markers in Hypogonadism
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Coskun Meric, MD, Gulhane School of Medicine
Other Study IDs: cmeric2000
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Hypogonadotropic Hypogonadism; Endothelial Dysfunction; Insulin Resistance
Keywords: Hypogonadism; Asymmetric Dimethyl Arginine; Osteoprotegerin; Fibroblast Growth Factor; Vitamin D
MeSH Terms: conditions — Hypogonadism; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control patients: BMI and age matched healthy male subjects
- hypogonadism patients: unconfounded group of patients with hypogonadism

SUMMARY:
The aim of this study is to investigate the markers of bone mineral metabolism in an unconfounded group of patients with hypogonadism and to search for a relationship between endothelial dysfunction and insulin resistance.

DETAILED DESCRIPTION:
Cardiometabolic disorders are prevalent in patients with hypogonadism. Endothelial dysfunction and insulin resistance are used in determining cardiovascular risk. The role of markers of bone mineral metabolism in hypogonadism is not clearly presented.

49 male patients with hypogonadotropic hypogonadism (HH) and 43 BMI and age matched healthy male subjects were enrolled. Osteoprotegerin (OPG), fibroblast growth factor-23 (FGF-23), vitamin D and asymmetric dimethylarginine (ADMA) levels were measured. The insulin sensitivity was estimated by homeostatic model assessment-insulin resistance (HOMA-IR) formula.

ELIGIBILITY:
Inclusion Criteria:

* male patients with hypogonadotropic hypogonadism
* being under the age of 45 and over the age of 18
* not previously given testosterone or human chorionic gonadotropin therapy
* not have any chronic metabolic disorders or organ dysfunction

Exclusion Criteria:

* female patients
* Other reasons hipogondism
* receive any treatment of hypogonadism
* presence of comorbid diseases

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study group was selected from the male subjects with hypogonadotropic hypogonadism who were not previously given testosterone or human chorionic gonadotropin therapy. The patients did not have any chronic metabolic disorders or organ dysfunction. Forty three age and BMI matched male volunteers were enrolled as control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Osteoprotegerin, Fibroblast Growth Factor 23 and Vitamin D3 levels | one year
  investigate the markers of bone mineral metabolism in patients with hypogonadism

SECONDARY OUTCOMES:
relationship between bone mineral metabolism and endothelial dysfunction, insulin resistance | one year

CONTACTS AND LOCATIONS:
Overall Officials: Coskun Meric, Principal Investigator — Gulhane School of Medicine Department of Endocrinology
Locations (1):
- Gulhane School of Medicine, Ankara, Turkey (Türkiye)